CLINICAL TRIAL: NCT06256107
Title: Exploring the Use of Virtual Reality Applications in Patients With a Diagnosis of Motor Neurone Disease
Brief Title: Virtual Reality in Motor Neurone Disease
Acronym: VR in MND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancashire Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 274505
Record Dates: First submitted 2022-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Motor Neuron Disease
MeSH Terms: conditions — Motor Neuron Disease

STUDY DESIGN:
Intervention Model Description: Device Feasibility
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention period will last 4 weeks where participants will be required to use the VR set and document the time of use in a daily diary
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — Virtual Reality Headset

SUMMARY:
Motor Neurone Disease (MND) is a chronic progressive neurological condition where people experience weakness of muscles leading to pain and restriction of movement as well as problems with swallowing, breathing and communication. The purpose of this study is to establish if Virtual Reality is useful for people with MND and if it helps improve their well being.

DETAILED DESCRIPTION:
Motor Neurone Disease (MND) is a chronic progressive neurological condition where people experience weakness of muscles leading to pain and restriction of movement as well as problems with swallowing, breathing and communication.

As people become increasingly immobile, they become restricted in their ability to perform activities of daily living, access the outdoors, participate in preferred occupational roles or engage in leisure activities. Consequently, there is a deterioration in their ability to experience well being and have quality of life. There is also a significant carer burden as the carer spends long hours in the day looking after the person. The average disease trajectory lasts between 3-5 years, followed by death. More recently, the use of Virtual Reality (VR) technology is being recognised in the field of health. This technology uses the interactions between an individual and a computer generated environment to stimulate different sensory modalities such as visual and auditory. The technology can be accessed commonly using head mounted goggles or head sets. The entertaining or stimulating effect of VR is useful in redirecting the person's attention away from the distressing experiences, such as pain and anxiety. The purpose of this study is to establish if VR is useful for people with MND and if it helps improve their well being.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MND
2. Sufficient cognitive ability to understand instructions with regards using the VR kit (ECAS score - minimum 100/136)
3. Has sufficient motor ability/dexterity to use the kit or a carer who will be able to assist with the use of the kit.
4. Can tolerate light and have sufficient head control to wear the head set.
5. English speaking

Exclusion Criteria:

1. Poor cognition - inability to understand instructions regarding the use of VR (Total ECAS Score <100/136)
2. Unable to tolerate light/unable to wear the head set
3. Light sensitive epilepsy, severe vertigo or dizziness.
4. Non English speaking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Edinburgh Mental Well being Scale | 4 weeks
  Quality of Life (Scale 0-10 higher being better)

SECONDARY OUTCOMES:
ECAS (Edinburgh Cognition Assessment Scale) | 4 weeks
  Cognition measure scale varied per question (Scale 0-8, 0-10, 0-12 higher being better)
PHQ-9 | 4 weeks
  scale for depression (Scale 0-27 - higher being worse)
GAD-7 | 4 weeks
  scale for anxiety (Scale 0-3 where higher is worse outcome)
ALS-FRS | 4 weeks
  test of function (Yes or No - ability to perform function)

CONTACTS AND LOCATIONS:
Overall Officials: Malabika Ghosh, PhD, Principal Investigator — Lancashire Teaching Hospitals NHS Foundation Trust
Locations (1):
- Lancashire Teaching Hospitals NHS Foundation Trust, Preston, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

DOCUMENTS (1):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT06256107/Prot_000.pdf